CLINICAL TRIAL: NCT07382388
Title: A Real-World Study on the Impact of Weight Loss on Treatment Efficacy in Overweight/Obese Patients With Plaque Psoriasis
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Guo Jin-Zhu, associate chief physician, Peking University Third Hospital
Other Study IDs: M20260001
Record Dates: First submitted 2026-01-20; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Weight Loss Group: receiving standard psoriasis care plus a personalized weight management program
  Interventions: Combination Product: Weight loss and psoriasis treatment
- Control Group: receiving standard psoriasis care only
  Interventions: Combination Product: psoriasis treatment

INTERVENTIONS:
Combination Product: Weight loss and psoriasis treatment — In the weight loss group, receive standardized treatment for their psoriasis based on disease severity and follow a personalized weight management plan, which may include dietary counseling, a tailored exercise regimen, and/or GLP-1 receptor agonist therapy (e.g., Semaglutide, Tirzepatide) if indicated.
  Groups: Weight Loss Group
Combination Product: psoriasis treatment — Receive standardized treatment for their psoriasis based on disease severity.
  Groups: Control Group

SUMMARY:
The goal of this investigator-initiated, real-world, observational study is to investigate the impact of weight loss on treatment efficacy in overweight or obese Chinese patients with moderate-to-severe plaque psoriasis.

The main question it aims to answer is:

Does a structured weight loss intervention (including dietary management, exercise, and/or pharmacotherapy) improve the clinical response to psoriasis therapy in this population, as measured by the proportion of patients achieving a Psoriasis Area and Severity Index (PASI) score below 3 at Week 24?

Researchers will compare the Weight Loss Intervention Group (receiving standard psoriasis care plus a personalized weight management program) to the Control Group (receiving standard psoriasis care only) to see if the addition of weight loss strategies leads to superior improvements in psoriasis severity, metabolic parameters, and quality of life.

Participants will:

Receive standardized treatment for their psoriasis based on disease severity.

Be allocated (based on patient preference and clinical judgment) to either the intervention or control group.

In the intervention group, receive and follow a personalized weight management plan, which may include dietary counseling, a tailored exercise regimen, and/or Glucagon-Like Peptide-1（GLP-1） receptor agonist therapy (e.g., Semaglutide, Tirzepatide) if indicated.

Undergo scheduled assessments at baseline, Week 12, and Week 24, including:

Clinical evaluations (PASI, Physician's Global Assessment, body surface area).

Anthropometric measurements (weight, BMI, waist/hip circumference).

Quality of life assessment (Dermatology Life Quality Index).

Safety monitoring for adverse events. To investigate the impact of weight loss on treatment efficacy among overweight/obese Chinese patients with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, regardless of gender.
2. Having signed the informed consent form.
3. Clinical diagnosis of plaque psoriasis.
4. Body Mass Index (BMI) categorized as overweight or obese.
5. For female patients: No plans for pregnancy or oocyte donation during the study period and voluntary use of highly effective physical contraception.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Individuals deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical diagnosis of plaque psoriasis and Body Mass Index (BMI) categorized as overweight or obese.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of PASI<3 at Week 24 | Week 24
  Proportion of patients undergoing weight loss treatment who achieve a Psoriasis Area and Severity Index (PASI) score below 3 at Week 24.

SECONDARY OUTCOMES:
Proportion of PASI<3 at Week 12 | Week 12
  Proportion of patients undergoing weight loss treatment who achieve a PASI score below 3 at Week 12.
Changes of BMI | Week 12 and Week 24
  Changes from baseline in Body Mass Index (BMI) at Week 12 and Week 24 in patients undergoing weight loss treatment.
Proportion of PGA 0/1 (Physician's Global Assessment) | Week 12 and Week 24
  Proportion of patients undergoing weight loss treatment who achieve a Physician's Global Assessment (PGA) score of 0 or 1 at Week 12 and Week 24.
Proportion of DLQI<6 | Week 12 and Week 24
  Proportion of patients undergoing weight loss treatment who achieve a Dermatology Life Quality Index (DLQI) score below 6 at Week 12 and Week 24